CLINICAL TRIAL: NCT01136889
Title: A Feasibility Study for a Randomised Controlled Trial of Pelvic Floor Muscle Training Combined With Vaginal Pessary for Women With Pelvic Organ Prolapse.
Brief Title: PEssary Plus Physiotherapy for Pelvic Organ Prolapse (PEPPY)
Acronym: PEPPY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glasgow Caledonian University (Other)
Collaborators: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Professor Suzanne Hagen, Nursing, Midwifery and Allied Health Professions (NMAHP) Research Unit
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RG957; Wellbeing of Women (Other: RG957); MREC (Other: Ref Number 07/S0703/141); NHS GG&C (Other: RO60139)
Record Dates: First submitted 2010-06-02; First posted 2010-06-04 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2011-01

CONDITIONS: Pelvic Organ Prolapse
Keywords: PFMT; Vaginal pessary; Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PFMT plus routine pessary management (Active Comparator): Women allocated to the intervention group will be invited to attend 5 out-patient appointments over a 16 week period with a trained specialist women's health physiotherapist at the study centre. Women will be taught how to contract the muscles, and also how to contract and hold prior to an event that increases intra-abdominal pressure ("the Knack"). Tailored advice will be given on ways of reducing intra-abdominal pressure, e.g. advice on weight loss, chronic cough, heavy lifting and general exercise. A prolapse specific Lifestyle Advice sheet will also be given to the women by the physiotherapist.
  Interventions: Other: PFMT
- Lifestyle (Active Comparator): Women allocated to the control group will be sent a Lifestyle Advice Leaflet only. They will have no planned intervention after their pessary is fitted, other than routine pessary management according to local protocols. The Lifestyle Advice Leaflet gives instructions on seeking advice, where appropriate, about weight loss, constipation, and avoidance of heavy lifting, coughing and high impact exercise, with a view to minimising increases in intra-abdominal pressure which may cause the prolapse to worsen.
  Interventions: Other: PFMT

INTERVENTIONS:
Other: PFMT — Women who have been successfully fitted with a vaginal pessary will be asked to attend five outpatient appointments over a 16 week period with a trained specialist women's health physiotherapist.
  Other Names: Pelvic Floor Muscle Training

SUMMARY:
1. To determine the feasibility of conducting a randomised controlled trial (RCT) of the effectiveness of a PFMT intervention in conjunction with vaginal pessary management versus vaginal pessary management alone for women with pelvic organ prolapse.
2. To develop and test the methods for a main trial.

The ultimate aim of a large multi-centre RCT would be to answer the question:

Is conservative management of pelvic organ prolapse with an individualised PFMT intervention in conjunction with vaginal pessary more effective than vaginal pessary alone in reducing prolapse-specific symptoms, prolapse severity and the need for further prolapse treatment?

DETAILED DESCRIPTION:
It is hypothesised that undertaking PFMT with a pessary in place may increase the level of existing muscle support in the pelvic area: by reducing the descent of the pelvic organs and the consequent stretching of soft tissue the pessary may allow the pelvic floor muscles to be exercised and strengthened more effectively. Potentially this could lead to additional improvements in the pessary retention rate and associated prolapse symptoms beyond that expected from the pessary alone. Urine, bowel and sexual function, which can be affected by prolapse, may also improve independently in response to a PFMT intervention. If a more permanent reduction in prolapse symptoms results from concurrent use of PFMT, this may delay or prevent the need for long term pessary use or surgical intervention. In summary, a PFMT intervention in combination with pessary management for vaginal prolapse may be more effective in reducing symptoms and increasing quality of life than management of the prolapse with a pessary alone. This study will start to provide the evidence to address this question.

This is a feasibility study to develop the methods for a multi-centre RCT. It will run alongside The POPPY Trial (a 17 centre trial of PFMT already underway in the UK; ClinicalTrials Number NCT00476892). Three of The POPPY Trial centres will be involved in this feasibility study. Over a 12 month period, we plan to enrol 50 women with diagnosed prolapse of stage I to IV, who are not eligible for The POPPY Trial because they require a pessary. These women will be randomised into one of two groups: PFMT (delivered by a physiotherapist at 5 appointments over 16 weeks) in conjunction with pessary management of their prolapse or pessary management alone. All women will have a nurse appointment six months after randomisation at which time their pessary will be removed. A replacement pessary will not be immediately re-fitted. At seven months after randomisation all women will have a review appointment with their gynaecologist to have their prolapse assessed, the pessary re-fitted if necessary, and other treatment needs discussed. Women will complete postal questionnaires, at baseline (prior to randomisation), at six months post-randomisation (prior to seeing the nurse to have the pessary removed), and seven months post-randomisation (prior to the 7 month gynaecologist review appointment), and record symptoms in a diary for one month after removal of the pessary. Key outcomes are: prolapse symptoms, prolapse-related quality of life, prolapse severity, and additional prolapse treatment received up to seven months after study entry.

ELIGIBILITY:
Inclusion Criteria:

Women:

* who are new attendees at outpatient gynaecology clinics with a primary complaint of prolapse;
* who have a prolapse of stage I to IV confirmed by their gynaecologist using the POP-Q grading system;
* who have a prolapse of one or more of the following types:
* anterior vaginal wall prolapse (urethrocele, cystocele,paravaginal defect);
* uterine/cervical prolapse;
* vaginal vault (after hysterectomy)prolapse;
* posterior vaginal wall prolapse (enterocele, rectocele, perineal deficiency);
* who require a vaginal pessary for treatment of their prolapse (the process of fitting the pessary will be according to standard practice at the centre thus the protocol for choice of pessary, insertion and follow-up will be determined locally);
* who successfully retain the vaginal pessary for two weeks after fitting;
* who are willing to participate in the study and to comply with their group allocation.

Exclusion Criteria:

Women:

* who wish surgical treatment for prolapse and wish to be immediately added to the surgical waiting list;
* who have had previous surgical treatment for prolapse;
* who have had a pessary fitted for treatment of prolapse within the last 12 months;
* who have had previous formal instruction in PFMT;
* who present with contraindications to either pessary or PFMT treatment;
* who are unable to comply with PFMT treatment;
* who have local atrophy (this must be treated first);
* who are less than 6-months postnatal;
* who are pregnant;
* who are unable to give informed consent.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-04; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Prolapse symptom score (POP-SS) | 7 months

SECONDARY OUTCOMES:
Prolapse-related quality of life(single item scored 0 to 10) | 7 months
Prolapse severity (POP-Q) | 7 months
Urinary, bowel and sexual symptoms | 7 months
Lifestyle changes | 7 months
General Health Status | 7 months
Recurrence of prolapse symptoms over the one month period between removal of the pessary (month 6) and gynaecology clinic review (month 7) | 7 months
Time without pessary (i.e. time from removal of pessary to pessary being re-fitted) | 7 months
Need for further prolapse treatment including continuing use of pessary, PFMT or surgery. | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Professor Suzanne Hagen, Principal Investigator — NMAHP Research Unit
Locations (4):
- United Kingdom (4):
  - Aberdeen Royal Infirmary, Aberdeen
  - Falkirk and District Royal Infirmary, Falkirk
  - Southern General Hospital, Glasgow
  - Victoria Infirmary, Glasgow

REFERENCES:
- [Derived] Bugge C, Adams EJ, Gopinath D, Stewart F, Dembinsky M, Sobiesuo P, Kearney R. Pessaries (mechanical devices) for managing pelvic organ prolapse in women. Cochrane Database Syst Rev. 2020 Nov 18;11(11):CD004010. doi: 10.1002/14651858.CD004010.pub4. PMID 33207004
- [Derived] Bugge C, Williams B, Hagen S, Logan J, Glazener C, Pringle S, Sinclair L. A process for Decision-making after Pilot and feasibility Trials (ADePT): development following a feasibility study of a complex intervention for pelvic organ prolapse. Trials. 2013 Oct 25;14:353. doi: 10.1186/1745-6215-14-353. PMID 24160371